CLINICAL TRIAL: NCT02466815
Title: Open-Label, Randomized, 3-Way Crossover Design to Assess the Relative Bioavailability of JNJ-42756493 Tablets
Brief Title: A Study to Assess the Relative Bioavailability of JNJ-42756493 Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CR107460; 42756493EDI1004 (Other: Janssen Research & Development, LLC); 2015-001583-19 (EudraCT Number)
Record Dates: First submitted 2015-06-05; First posted 2015-06-09 (Estimated); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Healthy
Keywords: Healthy; JNJ-42756493

ARMS (6):
- Treatment A, then Treatment B and then Treatment C (Experimental): Participants will receive treatment A (JNJ-42756493 10 milligram [mg] tablet, current clinical formulation [G-018] which uses milled active pharmaceutical ingredient [API]) in period 1, treatment B (JNJ-42756493 10 mg tablet, Prototype Formulation I [G-025] which uses coarser API) in period 2 and then treatment C (JNJ-42756493 10 mg tablet, Prototype Formulation II [G-025] which uses coarser API) in period 3.
  Interventions: Drug: JNJ-42756493 Current Clinical Formulation (G-018); Drug: JNJ-42756493 Prototype Formulation I (G-025); Drug: JNJ-42756493 Prototype Formulation II (G-025)
- Treatment B, then Treatment C and then Treatment A (Experimental): Participants will receive treatment B in period 1, treatment C in period 2 and then treatment A in period 3.
  Interventions: Drug: JNJ-42756493 Current Clinical Formulation (G-018); Drug: JNJ-42756493 Prototype Formulation I (G-025); Drug: JNJ-42756493 Prototype Formulation II (G-025)
- Treatment C, then Treatment A and then Treatment B (Experimental): Participants will receive treatment C in period 1, treatment A in period 2 and then treatment B in period 3.
  Interventions: Drug: JNJ-42756493 Current Clinical Formulation (G-018); Drug: JNJ-42756493 Prototype Formulation I (G-025); Drug: JNJ-42756493 Prototype Formulation II (G-025)
- Treatment A, then Treatment C and then Treatment B (Experimental): Participants will receive treatment A in period 1, treatment C in period 2 and then treatment B in period 3.
  Interventions: Drug: JNJ-42756493 Current Clinical Formulation (G-018); Drug: JNJ-42756493 Prototype Formulation I (G-025); Drug: JNJ-42756493 Prototype Formulation II (G-025)
- Treatment B, then Treatment A and then Treatment C (Experimental): Participants will receive treatment B in period 1, treatment A in period 2 and then treatment C in period 3.
  Interventions: Drug: JNJ-42756493 Current Clinical Formulation (G-018); Drug: JNJ-42756493 Prototype Formulation I (G-025); Drug: JNJ-42756493 Prototype Formulation II (G-025)
- Treatment C, then Treatment B and then Treatment A (Experimental): Participants will receive treatment C in period 1, treatment B in period 2 and then treatment A in period 3.
  Interventions: Drug: JNJ-42756493 Current Clinical Formulation (G-018); Drug: JNJ-42756493 Prototype Formulation I (G-025); Drug: JNJ-42756493 Prototype Formulation II (G-025)

INTERVENTIONS:
Drug: JNJ-42756493 Current Clinical Formulation (G-018) — JNJ-42756493 10 milligrams (2 tablets of 5 mg each) will be administered as current clinical formulation (G-018) in treatment A in either period 1, 2 or 3 as per treatment sequence.
Drug: JNJ-42756493 Prototype Formulation I (G-025) — JNJ-42756493 10 milligrams (2 tablets of 5 mg each) will be administered as Prototype Formulation I (G-025) in treatment B in either period 1, 2 or 3 as per treatment sequence.
Drug: JNJ-42756493 Prototype Formulation II (G-025) — JNJ-42756493 10 milligrams (2 tablets of 5 mg each) will be administered as Prototype Formulation II (G-025) in treatment C in either period 1, 2 or 3 as per treatment sequence.

SUMMARY:
The purpose of this study is to assess the relative bioavailability of 2 prototype G-025 tablets compared with the current G-018 tablet.

DETAILED DESCRIPTION:
This is an open-label (all people know the identity of the intervention), multi-period, randomized (study drug assigned by chance), single-dose, 3-way crossover study. The study consists of 21-day screening period, 3 open-label treatment periods with a minimum 21 (+-2)-day washout between doses, and end-of-study assessments 10 (+-2) days after the last dose. The duration of study is approximately 3 months. Participants will be randomized to 1 of 6 treatment sequences as follows: Treatment sequence 1=ABC, 2=BCA, 3=CAB, 4=ACB, 5=BAC AND 6=CBA. Treatment A=JNJ-42756493 current clinical formulation, 10 milligrams (mg) (2 tablets of 5 mg each). Treatment B= JNJ-42756493 Prototype Formulation I (G-025), 10 mg (2 tablets of 5 mg each) and Treatment C=JNJ-42756493 Prototype Formulation II (G-025), 10 mg (2 tablets of 5 mg each). Blood samples will be collected to determine pharmacokinetic parameters. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants should be willing to adhere to the prohibitions and restrictions specified in this protocol
* Woman must be either: postmenopausal (greater than (>) 45 years of age with amenorrhea for at least 2 years, or any age with amenorrhea for at least 6 months and a serum follicle stimulating hormone (follicle stimulating hormone [FSH]) >40 international unit per litre [IU/L]); surgically sterile
* Woman must have a negative serum beta-human chorionic gonadotropin (hCG) pregnancy test at screening and a negative urine pregnancy test on Day -1 of each treatment period
* Woman must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction during the study and for 3 months after receiving the last dose of study drug.
* Man who is sexually active with a woman of childbearing potential and has not had a vasectomy, must agree to use a highly effective method of contraception as deemed appropriate by the investigator and to not donate sperm during the study and for 3 months after receiving the last dose of study drug

Exclusion Criteria:

* Participants with history of or current clinically significant medical illness including (but not limited to) cardiac arrhythmias or other cardiac disease, hematologic disease, coagulation disorders (including any abnormal bleeding or blood dyscrasias), lipid abnormalities, significant pulmonary disease, including bronchospastic respiratory disease, diabetes mellitus, hepatic or renal insufficiency, thyroid disease, neurologic or psychiatric disease, infection, or any other illness that the investigator considers should exclude the subject or that could interfere with the interpretation of the study results
* Participants with history or current evidence of ophthalmic disorder, such as central serous retinopathy or retinal vein occlusion, active wet age related macular degeneration, diabetic retinopathy with macular edema, uncontrolled glaucoma, corneal pathology such as keratitis, keratoconjunctivitis, keratopathy, corneal abrasion, inflammation or ulceration
* Participants with clinically significant abnormal values for hematology, clinical chemistry, or urinalysis at screening or at Day -1 of Period 1 as deemed appropriate by the investigator
* Participants with clinically significant abnormal physical examination, vital signs, or 12-lead electrocardiogram (ECG) at screening or at Day -1 of Period 1 as deemed appropriate by the investigator
* Participants with use of any prescription or nonprescription medication (including vitamins and herbal supplements), except for paracetamol and hormonal replacement therapy within 14 days before the first dose of the study drug is scheduled until completion of the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2015-06; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of JNJ-42756493 | Predose, 0.16 hour (hr),0.33, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12 hr post-dose on Day 1; 24 and 36 hr post-dose on Day 2; 48hr post-dose on Day 3; 72hr post-dose on Day 4; 96hr post-dose on Day 5; 120hr post-dose on Day 6; 144hr post-dose on Day 7
  The Cmax is the maximum observed plasma JNJ-42756493 concentration. Relative bioavailability will be calculated by Cmax based on total drug concentrations.
Area Under the Plasma Concentration-time Curve From Time 0 to 24 Hours (AUC[0-24]) of JNJ-42756493 | Predose, 0.16 hour (hr),0.33, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12 hr post-dose on Day 1; 24 and 36 hr post-dose on Day 2; 48hr post-dose on Day 3; 72hr post-dose on Day 4; 96hr post-dose on Day 5; 120hr post-dose on Day 6; 144hr post-dose on Day 7
  AUC(0-24) is the area under the plasma JNJ-42756493 concentration-time curve from time 0 to 24 hours. Relative bioavailability will be calculated by AUC(0-24) based on total drug concentrations.
Area Under the Plasma Concentration-time Curve From Time 0 to Time of the Last Observed Quantifiable Concentration (Clast) (AUC[0-last]) of JNJ-42756493 | Predose, 0.16 hour (hr),0.33, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12 hr post-dose on Day 1; 24 and 36 hr post-dose on Day 2; 48hr post-dose on Day 3; 72hr post-dose on Day 4; 96hr post-dose on Day 5; 120hr post-dose on Day 6; 144hr post-dose on Day 7
  AUC(0-last) is the area under the plasma JNJ-42756493 concentration-time curve from time 0 to time of the last observed quantifiable concentration (Clast). Relative bioavailability will be calculated by AUC(0-last) based on total drug concentrations.
Area Under the Plasma Concentration-time Curve From Time 0 to Infinite Time AUC (infinity) of JNJ-42756493 | Predose, 0.16 hour (hr),0.33, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12 hr post-dose on Day 1; 24 and 36 hr post-dose on Day 2; 48hr post-dose on Day 3; 72hr post-dose on Day 4; 96hr post-dose on Day 5; 120hr post-dose on Day 6; 144hr post-dose on Day 7
  AUC (infinity) is the area under the plasma JNJ-42756493 concentration-time curve from time 0 to infinite time, calculated as the sum of AUC(0-last) and Clast/lambda(z), in which lambda(z) is the first-order rate constant associated with the terminal portion of the curve. Relative bioavailability will be calculated by AUC (infinity) based on total drug concentrations.

SECONDARY OUTCOMES:
Number of Participants With Adverse Events (AEs) or Serious Adverse Events (SAEs) | Screening up to end of study (up to 3 months)
  An AE is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; lifethreatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Merksem, Belgium